CLINICAL TRIAL: NCT06487871
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Effect of Fucoidan on Prostate Health in Males With Benign Prostatic Hyperplasia
Brief Title: A Study to Assess the Effect of Fucoidan on Prostate Health in Males With Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MN/231202/IP/BPH
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fucoidan extracted from Undaria pinnatifida (UPF) (Active Comparator): Two capsules to be taken after breakfast daily, with 200 ml glass of water for 90 days.
  Interventions: Dietary Supplement: Fucoidan extracted from Undaria pinnatifida (UPF)
- Placebo (Placebo Comparator): Two capsules to be taken after breakfast daily, with 200 ml glass of water for 90 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fucoidan extracted from Undaria pinnatifida (UPF) — Two capsules to be taken after breakfast daily, with 200 ml glass of water for 90 days.
  Arms: Fucoidan extracted from Undaria pinnatifida (UPF)
Dietary Supplement: Placebo — Two capsules to be taken after breakfast daily, with 200 ml glass of water for 90 days.
  Arms: Placebo

SUMMARY:
The present study is a randomized, double-blind, placebo-controlled study. Approximately 125 individuals will be screened, and considering a screening failure rate of 20%, at least 100 will be randomized in a ratio of 1:1 to receive either IP or placebo and will be assigned a unique randomization code. Each group will have not less than 40 completed participants after accounting for a dropout/withdrawal rate of 20%. The intervention duration for all the study participants is 90 days.

ELIGIBILITY:
Inclusion criteria:

* Males aged 45 to 80 years (inclusive of both ages) with a diagnosis of BPH established by a surgeon/nephrologist/urologist within the last 3 months and having any one of the two clinical as well as one of the radio-diagnostic parameters:-

  a) Clinical parameter: i) History of lower urinary tract symptoms ii) Rectal examination indicating increased prostate size. b) Radio-diagnostic parameter: i) Uroflowmetry (less than 20 ml/sec maximum flow rate [Qmax]) ii) Ultrasound Sonography (USG) - Enlargement of the central gland with a calculated urine volume exceeding 30 mL and increased post-micturition.
* Moderate symptoms with an IPSS Score more than or equal to 8-19.
* No signs of prostate cancer as indicated by 1-3 U/L of Prostatic Acid Phosphatase (PAP) in serum.
* Fasting blood glucose (FBG) less than 125 mg/dL.
* Willing to give voluntary written informed consent and adhere to all the requirements of the study.

Note: Only biological males will be included. During screening I, if participants are currently on drug/ supplement for BPH, a washout period of 10±2 days will be provided. After this period, the participant will be rescheduled for screening IA.

Exclusion Criteria:

* Males with no signs of inflammation as assessed by Erythrocyte Sedimentation Rate (ESR) of more than or equal to 20 mm/hr.
* Males with more than or equal to 3.5 ng/mL of PSA in serum.
* Males diagnosed with prostate cancer.
* Males who have recently started a bladder-training program within the last 30 days.
* Males who have undergone urogenital surgery.
* Males who have had a bladder biopsy and/or cystoscopy and biopsy within the last 30 days.
* Males who have had an indwelling catheter or practiced self-catheterization, and/or urethral stricture within the last 30 days.
* Males diagnosed with obstructive renal/urinary tract calculi.
* Males who have been medically diagnosed with chronic persistent local pathology (i.e., interstitial cystitis, prostatitis, etc.)
* Males with chronic inflammatory diseases such as Rheumatoid arthritis (RA), Ulcerative colitis, and Chronic obstructive pulmonary disease (COPD).
* Males receiving or prescribed anticoagulation therapy.
* Males who have been diagnosed with severe renal and/or hepatic insufficiency.
* Males who have been diagnosed with genital anatomical deformities.
* Males with a history of uncontrolled diabetes mellitus, uncontrolled hypertension (SBP/DBP ≥ 140/90 mmHg1 with or without medication), thyroid disorders, spinal cord injury, uncontrolled psychiatric disorder, and/or abnormal secondary sexual characteristics.
* Males who have a history of chronic alcohol (defined as consuming more than 5 drinks on any day or more than 15 drinks/week2) and/or illicit drug abuse.
* Males who have participated in any other clinical study during the last 30 days.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological males will be included.
Enrollment: 95 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
To assess the effect of Investigational product (IP) on prostate health as assessed by the International Prostate Symptom Score (IPSS) as compared to placebo. | Day 0
  The International Prostate Symptom Score (IPSS) consists of seven questions that assess both storage and voiding symptoms in participants with Benign Prostatic Hyperplasia (BPH).
  Respondents are presented with six response options for each of the seven questions, with scores ranging from 0 to 5 indicating the severity of the respective symptom. The total sum score, ranging from 0 to 35, aids in categorizing the severity of lower urinary tract symptoms (LUTSs): 0 - 7 indicates mild symptoms, 8 - 19 indicates moderate symptoms, and 20 - 35 indicates severe symptoms.
  Additionally, the final question of the IPSS addresses Quality of Life (QoL), with responses varying from "delighted" to "terrible" or scores from 0 to 6.
To assess the effect of Investigational product (IP) on prostate health as assessed by the International Prostate Symptom Score (IPSS) as compared to placebo. | Day 30
  The International Prostate Symptom Score (IPSS) consists of seven questions that assess both storage and voiding symptoms in participants with Benign Prostatic Hyperplasia (BPH).
  Respondents are presented with six response options for each of the seven questions, with scores ranging from 0 to 5 indicating the severity of the respective symptom. The total sum score, ranging from 0 to 35, aids in categorizing the severity of lower urinary tract symptoms (LUTSs): 0 - 7 indicates mild symptoms, 8 - 19 indicates moderate symptoms, and 20 - 35 indicates severe symptoms.
  Additionally, the final question of the IPSS addresses Quality of Life (QoL), with responses varying from "delighted" to "terrible" or scores from 0 to 6.
To assess the effect of Investigational product (IP) on prostate health as assessed by the International Prostate Symptom Score (IPSS) as compared to placebo. | Day 60
  The International Prostate Symptom Score (IPSS) consists of seven questions that assess both storage and voiding symptoms in participants with Benign Prostatic Hyperplasia (BPH).
  Respondents are presented with six response options for each of the seven questions, with scores ranging from 0 to 5 indicating the severity of the respective symptom. The total sum score, ranging from 0 to 35, aids in categorizing the severity of lower urinary tract symptoms (LUTSs): 0 - 7 indicates mild symptoms, 8 - 19 indicates moderate symptoms, and 20 - 35 indicates severe symptoms.
  Additionally, the final question of the IPSS addresses Quality of Life (QoL), with responses varying from "delighted" to "terrible" or scores from 0 to 6.
To assess the effect of Investigational product (IP) on prostate health as assessed by the International Prostate Symptom Score (IPSS) as compared to placebo. | Day 90
  The International Prostate Symptom Score (IPSS) consists of seven questions that assess both storage and voiding symptoms in participants with Benign Prostatic Hyperplasia (BPH).
  Respondents are presented with six response options for each of the seven questions, with scores ranging from 0 to 5 indicating the severity of the respective symptom. The total sum score, ranging from 0 to 35, aids in categorizing the severity of lower urinary tract symptoms (LUTSs): 0 - 7 indicates mild symptoms, 8 - 19 indicates moderate symptoms, and 20 - 35 indicates severe symptoms.
  Additionally, the final question of the IPSS addresses Quality of Life (QoL), with responses varying from "delighted" to "terrible" or scores from 0 to 6.

SECONDARY OUTCOMES:
To assess the effect of IP on urinary flow rate as assessed by uroflowmetry. | Day 0, Day 90
  Uroflowmetry is a simple procedure to assess urine flow rate over time. The machine provides results including maximum flow rate (Qmax), flow time, voided volume, and average flow rate. Typically, urine flow ranges from 10 ml to 21 ml per second. A low flow rate may indicate potential issues such as bladder neck or urethral obstruction or an enlarged prostate. Conversely, a high flow rate might suggest weak muscles surrounding the urethra or urinary incontinence problems.
To assess the effect of IP on Post void residual volume (PVR) as assessed by ultrasonography | Day 0, Day 90
  Post void residual volume (PVR) serves as a diagnostic indicator, representing the urine left in the bladder after voluntary voiding. The PVR measurement, typically obtained through a formal bladder ultrasound examination, precisely quantifies the remaining urine shortly after voiding.
  PVR volume of less than 50 mL is deemed sufficient for bladder emptying, while in the elderly, a range between 50 and 100 mL is considered normal. Typically, a PVR volume exceeding 200 mL is regarded as abnormal and may indicate incomplete bladder emptying or bladder outlet obstruction. A PVR volume surpassing 400 mL is considered high.
To assess the effect of IP on Prostate-specific antigen (PSA) in serum | Day 0, Day 90
  PSA, a kallikrein-like serine protease, is primarily produced by prostate epithelial cells to facilitate the liquefaction of ejaculate and support sperm motility. The standard PSA test measures total PSA, encompassing both bound (attached to proteins) and free (unbound) PSA. When both total PSA and free PSA levels are elevated, with a high percentage of free PSA, it typically indicates BPH rather than cancer.
To assess the effect of IP on Perceived immune status as assessed by Immune Status Questionnaire (ISQ) | Day 0, Day 30, Day 60, Day 90
  The ISQ is rated on a 5-point Likert scale from 0 to 4.The total sum of ISQ score ranges from 0 to 28, with higher scores indicating poorer immune status.

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - Sarjanam Hospital, Vadodara, Gujarat
  - NKP Salve Institute of Medical Science and Research Centre and Lata Mangeshkar Hospital, Nagpur, Maharashtra
  - Rising Medicare Hospital Name of, Pune, Maharashtra
  - Pawana Hospital, Pune, Maharashtra
  - Bhalerao Clinics, Pune, Maharashtra
  - Jaipur National University of Medical Science and Research Centre Name of, Jaipur, Rajasthan